CLINICAL TRIAL: NCT01166919
Title: Pilot Study on the Use of the Matrix Radiofrequency for Treatment of Port Wine Stain Birthmarks
Brief Title: Pilot Study on the Use of the Matrix Radiofrequencyfor Treatment of Port Wine Stain Birthmarks
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Laser company cannot provide laser unit for the study.
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J.S.Nelson, MD,PhD,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20097262
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medical Tool (Experimental): Matrix Radiofrequency Treatment of Port Wine Stain Birthmarks
  Interventions: Device: Matrix Radiofrequency

INTERVENTIONS:
Device: Matrix Radiofrequency — Matrix Radiofrequency Treatment of Port Wine Stain Birthmarks

SUMMARY:
Port wine stain, also called nevus flammeus, is a congenital, cutaneous vascular malformation involving post-capillary venules which produces a light pink to red to dark-red-violet discoloration of the skin. It is estimated that Port wine stain occurs in 3 children per 1,000 live births. Approximately 900,000 individuals in the United States and twenty million people worldwide have Port wine stain birthmarks .

DETAILED DESCRIPTION:
The purpose of this research study is to improve port wine stain treatment after Matrix Radiofrequency device treatment. The Matrix Radiofrequency device energy generates fractional deep dermal heating in the region of the electrode matrix to induce skin injury, thus eliciting a wound healing response. Less affected tissue surrounding the matrix points may be stimulated by heat which helps accelerate the healing process, while at the same time minimizing adverse effects such as scarring or changes in the normal skin pigmentation.

The researcher can determine Port wine stain areas treated with the Matrix Radiofrequency device will have improved Port wine stain blanching responses as compared to those areas treated by pulsed dye laser.

ELIGIBILITY:
Inclusion Criteria:

* Port Wine Stain Birthmarks suitable for comparison testing
* Age > 18 years of age

Exclusion Criteria:

* Less than 18 years old
* Are pregnant or breastfeeding
* Other history assess by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Medical Tool | 8 weeks
  Matrix Radiofrequency Treatment of Port Wine Stain Birthmarks

SECONDARY OUTCOMES:
Port Wine Stain blanching | 8 weeks
  Blanching responses on test site will be obtained from visible reflectance spectroscopy and Port Wine Stainblood volume fractions in the skin before and after laser treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Nelson, M.D,PhD, Principal Investigator — Beckman Laser Institute University of California Irvine